CLINICAL TRIAL: NCT06899412
Title: Clinical Evaluation of Success Rate of Deep Marginal Elevation Technique Using Self-adhesive Flowable Composite Versus Conventional Bonded Flowable Composite: Randomized Clinical Trial
Brief Title: Rct Deep Margin Elevation by Self Adhesive Composite
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Elsayed Ramadan, Dr.hadeer elsayed, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 14422023446877
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Deep Margin Elevation
Keywords: deep margin; composite restorations; class II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Active Comparator)
  Interventions: Other: Conventional flowable composite
- Group 2 (Experimental)
  Interventions: Other: self adhesive flowable composite

INTERVENTIONS:
Other: self adhesive flowable composite — FIT SA is a self-adhesive, light-cured, flowable restorative with two discrete viscosities, F03 (low flow) and F10 (high flow) UDMA,HEMA,Phosphonic acid monomer, S-PRG filler based on fluoroboroaluminosilicate glass, Polymerizationinitiator,Pigments and others, Shofu's exclusive GIOMER technology gives FIT SA the ability to release and recharge fluoride and other beneficial ions for the life of the restoration.
  Arms: Group 2
Other: Conventional flowable composite — Conventional flowable composite (bulk fil)
  Arms: Group 1

SUMMARY:
This study intend to study the development and introduction of new efficient approaches to overcome the problems of technique sensitivity of deep margin elevation by conventional flowable composite. This new class of Self- adhesive composites that have been developed and were marketed as flowable, low viscosity resin composites does not require any etching or bonding strategy before cavity filling and the ability to wet and adapt easily.The procedure is simplified by eliminating the adhesive application, which is the most technique sensitive step. (Fu J, Kakuda S, Pan F, e t al. 2013).

DME addresses multiple clinical problems associated with sub-gingival margins which pose a challenge due to limited access, rubber dam slippage over the margin and subsequent persistent saliva,

crevice fluid and blood leakage. There are uncertainties within the profession in providing DME, and it is still considered a new approach. A recent survey revealed 78% of dentists had more than one concern about the procedure, ranging from isolation and inspection, marginal adaptation, microleakage. (Taylor, Burns, 2024) FIT SA™, a new comprehensive self-adhesive flowable restorative with bioactive Giomer Technology inside. FIT SA has eliminated the need for the technique sensitive bonding procedure. FIT SA offers superior strength and polishability, and the unique filler structure combines the light transmission and diffusion properties of enamel and dentin to blend well withthe surrounding dentition.

DETAILED DESCRIPTION:
Deep margin elevation (DME), or coronal margin relocation (CMR), is a procedure used to raise or reposition sub-gingival margins into supra-gingival margins using several materials to increase marginal integrity and bonding strength. Dietschi and Spreafico proposed the DME technique in 1998 to solve the problems associated with sub-gingival restorations. Despite this fact, it is still considered a new approach. Nowadays, clinical dentistry is directed toward conservatism, where in several situations the minimally invasive DME can replace the invasive procedures of crown lengthening. Sub-gingival preparations present difficulties that may complicate all further steps, such as rubber dam isolation, impression taking both digitally and traditionally, placement of a restoration, cementation as well as cervical area finishing and polishing. Moreover, indirect partial posterior restorations often display sub- gingival margins, which are accompanied by both biological and operative problems. Operative problems are attributed to changes in the tooth structure that are associated with deep margins, such as the absence of enamel, where dentin and cementum will pose more difficulties in bonding. Up until now, there is a limitation in the studies assessing the advantages and limitations of DME, most of them are in vitro concentrating on fracture resistance, bond strength, and marginal adaptation of indirect restorations. (Aldakheel, Almuhtab et al.2022).

ELIGIBILITY:
Inclusion Criteria:

Patients accept the one year follow up period. Cooperative patients. The study recruited volunteers of both genders Age from 21 to 45 years Primary compound proximal caries, with International Caries Detection and Assessment System (ICDAS) scores of 4 or 5.

The buccolingual width of the lesion could not exceed two-thirds of the intercuspal distance.

The remaining dentin thickness not less than 1 mm from the pulp and that could be identified clinically and by periapical xray Vital teeth without any signs of radiolucency in the periapical or furcation areas.

Participants also had to present a moderate risk of caries.

Exclusion Criteria:

Those who requiring any form of pulp capping will excluded to differentiate postoperative hypersensitivity from pulpal inflammation.

Individuals with poor oral hygiene. Patients undergoing orthodontic treatment. Periodontal surgery patients. Smokers. Pregnant women. Patients without occlusal contact. Those suffering prolonged tooth pain that disrupted sleep.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
post operative hyper sensitivity | 1 year
  Patients will be recalled at 3, 6, and 12 month post treatment to assess the occurrence of POH by verbally questioning the patient regarding sensitivity to cold, hot, sweet stimuli, mastication and clenching. Their answers about presence and degree of severity in sensitivity were measured using Visual Analogue Scale (VAS). The VAS is presented as a 10 cm horizontal line anchored by two extremes, no pain (score 0) and pain as bad as it could be (score 10). Patients were asked to choose the mark that represented their degree of pain, which was assigned to be one of four categorical score: None; (0), Mild (1- 3), Moderate (4-6) and Severe (7-10). All the readings (marks) stated by the patients will be recorded and then the amount of pain will be assessed. Data will be collected, computerized and statistically analyzed using Medcalc software, version 22 for windows (MedCalc Software Ltd, Ostend, Belgium)